CLINICAL TRIAL: NCT02427724
Title: The Effect of Topical Anesthetic Using Lidocaine 2.5%/Prilocaine 2.5% Versus Lidocaine 7%/Tetracaine 7% Cream on Patients' Pain and Operative Experience During Treatment With QSwitched 532nm Laser
Brief Title: The Effect of Topical Anesthetics on Patients' Pain and Operative Experience During Treatment With QSwitched Laser
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STU200401
Record Dates: First submitted 2015-04-13; First posted 2015-04-28 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Lentigo
MeSH Terms: conditions — Lentigo | interventions — Lidocaine; Prilocaine; Anesthetics, Local; Tetracaine; Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- lidocaine 2.5%/prilocaine 2.5% topical anesthetic (Active Comparator): Subjects will be screened, assessed, and randomized to be treated with a single pass of the Q-switched 532nm laser after application of LPTA, LTTA, or PV under occlusion to the assigned randomized site.
  Interventions: Drug: lidocaine 2.5%/prilocaine 2.5% topical anesthetic; Device: Q-switched 532nm Laser
- lidocaine 7%/tetracaine 7% topical anesthetic (Active Comparator): Subjects will be screened, assessed, and randomized to be treated with a single pass of the Q-switched 532nm laser after application of LPTA, LTTA, or PV under occlusion to the assigned randomized site.
  Interventions: Drug: lidocaine 7%/tetracaine 7% topical anesthetic; Device: Q-switched 532nm Laser
- placebo vehicle (Placebo Comparator): Subjects will be screened, assessed, and randomized to be treated with a single pass of the Q-switched 532nm laser after application of LPTA, LTTA, or PV under occlusion to the assigned randomized site.
  Interventions: Drug: placebo vehicle; Device: Q-switched 532nm Laser

INTERVENTIONS:
Drug: lidocaine 2.5%/prilocaine 2.5% topical anesthetic
  Arms: lidocaine 2.5%/prilocaine 2.5% topical anesthetic
Drug: lidocaine 7%/tetracaine 7% topical anesthetic
  Arms: lidocaine 7%/tetracaine 7% topical anesthetic
Drug: placebo vehicle
  Arms: placebo vehicle
Device: Q-switched 532nm Laser

SUMMARY:
This study will conduct a split-face and -body randomized control trial to compare lidocaine 2.5%/prilocaine 2.5% topical anesthetic (LPTA), lidocaine 7%/tetracaine 7% topical anesthetic (LTTA), and placebo vechicle (PV) on patients' pain perceptions with Q-switched 532nm laser for the treatment of lentigines and/or photorejuvenation.Subjects will fill out a pain score on a visual analog scale (VAS) with 0 being no pain and 10 being most pain after each treatment area is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have moderate lentigines and/or photodamage and desire laser toning.
2. Females 25-65 years of age.
3. In good health.
4. Have Fitzpatrick phototype I-III.
5. Willingness and the ability to understand and provide informed consent and communicate with the investigator/study staff.

Exclusion Criteria:

1. Younger than 25 or older than 65 years of age.
2. Pregnant or lactating.
3. Is a male.
4. Has received the following treatments on the face:

   * ablative or non-ablative laser procedure in the past 3 months
   * radiofrequency device treatment in the past 3 months
   * ultrasound device treatment in the past 3 months
   * medium to deep chemical peel in the past 3 months
5. Has an active infection on the face or upper inner arms (excluding mild acne).
6. Is allergic to lidocaine, tetracaine, or prilocaine.
7. Has kidney disease and/or liver disease.
8. Has G-6-PD and/or pseudocholinesterase deficiency.
9. Is taking a class I anti-arrhythmic medication.
10. Is tanned.
11. Has a history of hyperpigmentation with laser treatment.
12. Has a mental illness.
13. Has a history of a chronic pain condition such as fibromyalgia or vulvodynia.
14. Unable to understand the protocol or to give informed consent.
15. Multiply recurrent episodes of cold sores.
16. Any significant skin disease beyond mild acne.
17. Any other condition that would, in the professional opinion of the investigator, potentially affect response or participation in the clinical clinical study, or would pose as an unacceptable risk to the subject.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-04; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
visual analog score (VAS) pain rating | Day of treatment
  Subjects will fill out a visual analog score (VAS) pain rating after treatment with 0 being no pain and 10 being worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States